CLINICAL TRIAL: NCT07366814
Title: Comparison of Pipelle and Karman Endometrial Biopsy Methods Under Standardized Paracervical Block: A Prospective Randomized Study
Brief Title: Pipelle Versus Karman Endometrial Biopsy Under Standardized Paracervical Block
Acronym: PB-EMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Betül Bacak, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EK-193-2025-EMB
Record Dates: First submitted 2026-01-03; First posted 2026-01-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Abnormal Uterine Bleeding; Postmenopausal Bleeding
Keywords: Endometrial Biopsy; Pipelle; Karman Cannula; Paracervical Block; Abnormal Uterine Bleeding; Postmenopausal Bleeding; Diagnostic Adequacy; Patient Satisfaction
MeSH Terms: conditions — Metrorrhagia; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Eligible participants are randomly assigned in a 1:1 ratio to undergo endometrial biopsy using either the Pipelle device or the Karman cannula, with both groups treated concurrently.
Who Masked: Outcomes Assessor
Masking Description: Histopathological evaluation of endometrial samples is performed by pathologists who are blinded to the biopsy method used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pipelle Endometrial Biopsy (Experimental): Participants assigned to this arm undergo office-based endometrial biopsy using a Pipelle device. All procedures are performed under standardized paracervical block anesthesia with the same anesthetic agent, dose, and technique as the other study arm.
  Interventions: Device: Pipelle Endometrial Biopsy
- Karman Endometrial Biopsy (Experimental): Participants assigned to this arm undergo office-based endometrial sampling using a Karman cannula. All procedures are performed under standardized paracervical block anesthesia with the same anesthetic agent, dose, and technique as the other study arm.
  Interventions: Device: Karman Cannula Endometrial Biopsy

INTERVENTIONS:
Device: Pipelle Endometrial Biopsy — Endometrial sampling performed using a Pipelle device in an outpatient setting. The procedure is conducted under standardized paracervical block anesthesia using the same anesthetic agent, dose, and technique for all participants.
  Other Names: Pipelle de Cornier
  Arms: Pipelle Endometrial Biopsy
Device: Karman Cannula Endometrial Biopsy — Endometrial sampling performed using a Karman cannula in an outpatient setting. The procedure is conducted under standardized paracervical block anesthesia using the same anesthetic agent, dose, and technique for all participants.
  Other Names: Karman Cannula; Manual Vacuum Aspiration Cannula
  Arms: Karman Endometrial Biopsy

SUMMARY:
Endometrial biopsy is a commonly used outpatient procedure to evaluate abnormal uterine bleeding and postmenopausal bleeding. Different sampling methods are available, but their diagnostic adequacy and patient experience may vary.

This prospective randomized study compares two commonly used endometrial biopsy methods, Pipelle and Karman cannula, under standardized paracervical block anesthesia. All participants receive the same local anesthetic technique to minimize pain-related differences between methods.

The primary objective is to compare the rate of clinically adequate endometrial samples obtained with each method. Secondary outcomes include patient-reported pain, patient satisfaction, procedure duration, need for additional diagnostic procedures, and hospital-related costs.

Study findings are expected to support clinical decision-making regarding the most effective and practical endometrial biopsy method when adequate pain control is provided.

DETAILED DESCRIPTION:
Endometrial biopsy is an essential diagnostic procedure in the evaluation of abnormal uterine bleeding and postmenopausal bleeding. Office-based endometrial sampling techniques are widely used because these techniques are minimally invasive and cost-effective; however, diagnostic adequacy, patient tolerance, and resource utilization may differ between methods.

Pain during the procedure is a major factor affecting patient experience and may confound comparisons between sampling techniques. To address this limitation, participants receive a standardized paracervical block using the same anesthetic agent, dose, and technique, allowing the comparison to focus on the intrinsic performance of the biopsy methods rather than differences in analgesia.

This is a prospective, randomized, parallel-group study. Eligible participants undergoing endometrial biopsy are randomly assigned in a 1:1 ratio to either Pipelle endometrial biopsy or Karman cannula endometrial sampling. Randomization is stratified by menopausal status. Procedures are performed in an outpatient setting according to routine clinical practice.

Histopathological evaluation of endometrial samples is performed by pathologists blinded to the sampling method. Sample adequacy is assessed based on predefined criteria, with a focus on whether the specimen provides sufficient information for clinical decision-making.

In addition to diagnostic adequacy, patient-reported outcomes, including pain and satisfaction with the procedure, are assessed. Procedure duration, need for additional diagnostic interventions due to inadequate sampling, and hospital-related costs associated with each method are also evaluated.

Standardized analgesia and inclusion of clinical, patient-centered, and economic outcomes are intended to provide practical evidence to guide the selection of endometrial biopsy methods in routine gynecologic practice.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 years or older
* Abnormal uterine bleeding or postmenopausal bleeding requiring endometrial sampling
* Ability to provide written informed consent
* Eligible for office-based endometrial biopsy

Exclusion Criteria:

* Pregnancy
* Active pelvic infection
* Known cervical or endometrial cancer
* Severe cervical stenosis preventing endometrial sampling
* Known bleeding disorders or use of anticoagulant therapy that contraindicates biopsy
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2026-01-03 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-02-09 (Actual)

PRIMARY OUTCOMES:
Clinically Adequate Endometrial Sample Rate | At the index procedure (same day)
  Proportion of endometrial biopsy samples considered clinically adequate for diagnosis based on blinded histopathological assessment.

SECONDARY OUTCOMES:
Procedure-Related Pain Score | Periprocedural
  Eligible participants undergo outpatient endometrial sampling under a standardized analgesia protocol: 3 mL of 2% prilocaine is injected for a paracervical block at the 1 and 11 o'clock positions before tenaculum application, followed by a 2-minute waiting period; a tenaculum is then applied and endometrial sampling is performed using either a Pipelle device or a 5-mm Karman cannula according to random assignment. Sampling is recorded as the number of predefined sampling cycles (maximum 3), and cervical stenosis, need for dilation, procedure duration, additional analgesia (e.g., NSAIDs), and complications are documented. Specimens are placed immediately in formalin in identical containers labeled with study ID only, sent daily in mixed order, and evaluated by pathologists blinded to sampling method for adequacy and diagnosis (including reason for inadequacy). Pain is assessed using the Visual Analog Scale for Pain (0-10; higher scores indicate worse pain) during the procedure and at 3
Patient Satisfaction With the Procedure | Same day after the procedure
  Patient-reported satisfaction with the endometrial biopsy procedure assessed using a Likert-type questionnaire, including willingness to undergo the same procedure again if needed.
Procedure Duration | During the procedure
  Time required to complete the endometrial biopsy procedure, measured from speculum insertion to completion of tissue sampling.
Need for Additional Diagnostic Procedures | Within 2 weeks after the procedure
  Proportion of participants requiring additional diagnostic procedures due to an inadequate endometrial biopsy sample.
Hospital-Related Cost per Participant | Within 2 weeks after the procedure
  Total hospital-related cost per participant, including procedural costs and costs related to additional diagnostic interventions when required.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ketenci Gencer, Assoc. Prof., Study Director — University of Health Sciences, Gaziosmanpaşa Training and Research Hospital
Locations (1):
- University of Health Sciences, Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to local ethical regulations and the need to protect participant privacy. The dataset contains sensitive clinical information, and no consent for public data sharing was obtained from participants.

REFERENCES:
- [Result] Coskun ES, Yeniocak AS, Bacak HB, Salman S. Optimizing analgesia for endometrial biopsy: A prospective, randomized comparative study. J Obstet Gynaecol Res. 2025 Jan;51(1):e16148. doi: 10.1111/jog.16148. Epub 2024 Nov 17. PMID 39551483